CLINICAL TRIAL: NCT02903420
Title: A Clinical Trial for Transcatheter Aortic Valve Implantation in Chronic Dialysis Patients With Aortic Valve Stenosis
Brief Title: A Clinical Trial of Transcatheter Aortic Valves in Dialysis Patients (Japan)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EW-P-003
Record Dates: First submitted 2016-08-22; First posted 2016-09-16 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SAPIEN 3 (Experimental): Transcatheter Aortic Valve Implantation (TAVI) with the Edwards SAPIEN 3 Transcatheter Heart Valve and Delivery System
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Implantation of Edwards SAPIEN 3 Transcatheter Heart Valve (Model: 9600TFX) via transfemoral, transapical or transaortic approach.

SUMMARY:
A single arm, prospective, open, non-randomized, Japanese multicenter trial to evaluate the safety and effectiveness of the Edwards SAPIEN 3 Transcatheter Heart Valve System (Model: 9600TFX) in the treatment of symptomatic severe aortic stenosis patients on chronic dialysis, who are determined by the heart team to be unable to undergo safe open surgical therapy and have the benefits of the study valve implantation. Following completion of enrollment, subjects will be eligible for enrollment in the continued access phase of the trial.

DETAILED DESCRIPTION:
1-year mortality after the study valve implantation will be compared to the performance goal based on the literature review of clinical outcomes for dialysis patients who underwent surgical aortic valve replacement. Data will be collected from all patients for up to five years following the index valve replacement procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is determined by the heart team to be unable to undergo open surgical therapy and have the benefits of the study valve implantation.
* Patient has senile degenerative aortic valve stenosis
* Patient has been on dialysis (hemodialysis or peritoneal dialysis) in stable condition for ≥ 3 months.
* Patient has appropriate aortic valve annulus size measured by TEE or 3D-CT.

Exclusion Criteria:

* Patient has evidence of an acute myocardial infarction (MI) within 30 days prior to the index procedure.
* Patient has a congenital unicuspid or bicuspid aortic valve, or non-calcified aortic valve.
* Patient has severe aortic valve regurgitation.
* Patient has severe mitral valve regurgitation.
* Patient has an experience of any therapeutic invasive cardiac procedures within 30 days prior to the index procedure. Implantation of a permanent pacemaker or balloon valvuloplasty for bridging to procedure after a qualifying echo are not considered exclusionary.
* Patient with planned concomitant surgical or transcatheter ablation for atrial fibrillation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2026-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiki Sawa, Principal Investigator — Osaka University Hospital
Locations (2):
- Japan (2):
  - Osaka University Hospital, Suita, Osaka
  - Keio University Hospital, Shinjuku-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-eight subjects were consented to the trial. Two subjects withdrawn from the study prior to the TAVI procedure. One subject had a gastrointestinal bleed prior to the procedure and the other subject had surgery per the decision of the surgeon.
Pre-assignment Details: Eight of the 36 subjects were treated as "bailout" due to the non-nominal volumes. The primary analysis was performed on the patients with nominal volume (n=28).
Period: Overall Study
Arm/Group | SAPIEN 3
Started | 28
Completed | 25
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 28
Region of Enrollment [Number; unit: participants]
  Japan | 28
Duration of Dialysis [Mean (Standard Deviation); unit: Years] — Dialysis is the process of removing excess water, solutes, and toxins from the blood in people whose kidneys can no longer perform these functions naturally.
  Years | 11.52 (10.47)
STS Score [Mean (Standard Deviation); unit: Units on a Scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  Units on a Scale | 14.34 (6.23)

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of Deaths
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 28
Participants | 3

2. Secondary Outcome: Device Success
Description: Number of patients with device success, defined as absence of procedural mortality, correct positioning of a study valve into the proper anatomical location, and intended performance of the study valve (no prosthesis-patient mismatch and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, and no moderate or severe prosthetic valve regurgitation).
Time Frame: 30 days
Population: Echo data was missing for one patient.
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 27
Participants | 20

3. Secondary Outcome: Hospitalization Length of Stay
Description: Discharge is defined as an average for 7 days
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 28
Days | 6.3 (2.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | SAPIEN 3
All-Cause Mortality (participants affected / at risk) | 3/28
Serious Adverse Events (participants affected / at risk) | 17/28
Other Adverse Events (participants affected / at risk) | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAPIEN 3 (N=28)
Angina pectoris (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Subarachnoid haematoma (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAPIEN 3 (N=28)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Atrioventricular block first degree (Cardiac disorders) | 2 (2)
Bundle branch block left (Cardiac disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 2 (2)
Shunt stenosis (Injury, poisoning and procedural complications) | 4 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Without the Sponsor's prior written consent, the Principal Investigator shall not publish the clinical study results or any documents containing any Study information at any academic conferences or in any publications of any nature.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT02903420/Prot_SAP_000.pdf